CLINICAL TRIAL: NCT06365463
Title: Telerehabilitation to Improve Balance and Mobility in Patients After Stroke: Group Physiotherapy Performed in Individuals' Homes
Brief Title: Telerehabilitation to Improve Balance and Mobility in Patients After Stroke
Acronym: TeleHome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: URIS202401
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Hemorrhagic Stroke; Ischemic Stroke
Keywords: Stroke; Telerehabilitation; Balance; Mobility
MeSH Terms: conditions — Hemorrhagic Stroke; Ischemic Stroke; Stroke | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telerehabilitation group (Experimental): Remote group training to improve balance and mobility
  Interventions: Behavioral: Telerehabilitation

INTERVENTIONS:
Behavioral: Telerehabilitation — The training will last for 6 weeks, with two 60-minute sessions of balance and mobility training per week. Two consecutive groups will participate.

SUMMARY:
Telerehabilitation is an effective rehabilitation method that allows patients to receive physiotherapy remotely in their homes. The purpose of this study was to investigate the effects of home-based remote group training for balance and mobility on activities and body functions.

DETAILED DESCRIPTION:
Patients in the chronic post-stroke phase will be assessed for balance and mobility before and after remotely conducted group training. The training will last for 6 weeks, with two 60-minute sessions of balance and mobility training per week. Two consecutive groups will participate. The participants's balance and weight-bearing symmetry will be comprehensive assessed, as well their sit-to-stand ability, walking speed, and satisfaction with the remote training. Detailed inclusion and exclusion criteria are specified in the appropriate section.

ELIGIBILITY:
Inclusion Criteria:

* chronic phase of ischemic or haemorrhagic stroke (>6 months after stroke)
* ability to walk independently on level ground or on all surfaces with or without a walking aid
* mild balance deficit
* sufficient cognitive and communicative abilities for participation
* access to a personal computer with a camera, connected to the Internet

Exclusion Criteria:

* stroke in the brainstem or cerebellum
* additional neurological condition
* musculoskeletal impairments that would interfere with the training
* advanced heart failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Change in balance | Assessment 1-5 days before and 1-5 days after the training
  Assessed using Mini-Balance Evaluation Systems Test (scale score range 0-28; higher scores mean a better outcome)
Change in limits of stability | Assessment 1-5 days before and 1-5 days after the training
  Assessed using a force plate
Change in weight-bearing symmetry | Assessment 1-5 days before and 1-5 days after the training
  Assessed using a force plate

SECONDARY OUTCOMES:
Change in mobility | Assessment 1-5 days before and 1-5 days after the training
  Assessed using 5 Times Sit-to-Stand test (measured in seconds; longer times a worse outcome)
Change in walking speed | Assessment 1-5 days before and 1-5 days after the training
  Assessed using 10-Meter Walk Test (expressed in metres/second; higher speed means a better outcome)

OTHER OUTCOMES:
Satisfaction with the remote training | Assessed 1-5 days after the training
  Assessed using the Modified Physical Activity Enjoyment Scale (scale score expressed as percentage; higher scores mean a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Urška Puh, PT, PhD, Principal Investigator — University Rehabilitation Institute, Rehabilitation of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia